CLINICAL TRIAL: NCT06317844
Title: Examination of Psychological and Physiological Pathways Linking Gratitude and Pain and the Moderating Effects of COMT Genotype on These Associations
Brief Title: Examination of Psychological and Physiological Pathways Linking Gratitude and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BlackHillsHealthPsych; P20GM103443 (NIH)
Record Dates: First submitted 2024-03-06; First posted 2024-03-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Pain; Positive Thinking; Emotions
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude Writing (Experimental): In the gratitude writing condition, participants will write continuously for 5 minutes about someone they are grateful for.
  Interventions: Behavioral: Behavioral Writing Intervention
- Neutral Writing (Placebo Comparator): Participants in the neutral writing condition will write continuously for 5 minutes about how they got to the research laboratory.
  Interventions: Behavioral: Behavioral Writing Intervention

INTERVENTIONS:
Behavioral: Behavioral Writing Intervention — This behavioral intervention will require participants to write about certain aspects of their lives.

SUMMARY:
The goal of this clinical trial is to compare the effects of a brief gratitude intervention on individuals' psychological and physiological responses to acute pain. Furthermore, these associations will be examined in the context of genetic variations associated with both pain and psychological processes.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be randomized to a behavioral writing intervention and a cold pressor task. Participants will be randomized to a gratitude or neutral writing condition.

ELIGIBILITY:
Inclusion Criteria:

* must be pain-free
* must be at least 18 years old

Exclusion Criteria:

* cardiovascular disease
* Raynaud's disease
* epilepsy
* being pregnant
* having a current injury to or open cut or sore on one's non-dominant hand
* history of fainting or seizures
* history of frostbite in non-dominant hand
* chronic pain conditions (e.g., fibromyalgia, neuropathy, arthritis)
* diabetes
* malignant tumor
* chronic lung disease
* liver disease
* kidney disease
* gastrointestinal diseases
* currently taking opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Pain Ratings from Baseline to 10-minutes Post Cold Pressor Test | Baseline to 10 minutes post cold pressor test
  Self-reported measures of pain will be reported on a numeric scale of 0 (no pain) to 10 (strongest pain imaginable every 15 seconds throughout a cold pressor test and again 1 minute and 10 minutes post cold pressor test.
Differences in Pain Tolerance to Cold Pressor Test | Up to 1.5 minutes of Cold Pressor Test
  Pain tolerance will be measured in terms of how many seconds individuals can keep their hand submerged in near-freezing water, for a maximum of up to 90 seconds (the task will be ended at that point).
Differences in Pain Onset to Cold Pressor Test | Up to 1.5 minutes of Cold Pressor Test
  Pain onset will be measured in seconds between participants submerging their hands into near-freezing water and the self-reported beginning of pain.

SECONDARY OUTCOMES:
Differences in Pain-Related Cognition | Immediately after the Cold Pressor Test
  The Rumination and Reappraisal subscales from the Pain-Related Cognitive Processes Questionnaire will be used to assess the extent to which individuals engaged in various thought processes during the cold pressor test. Each subscale is comprised of 6-items and answered on a 0 (Not at all) to 4 (All or most of the time) scale.
Differences in Autonomic Nervous System Responsivity | Baseline to 10 minutes post cold pressor test
  Autonomic nervous system responsivity will be assessed using levels of salivary alpha-amylase. Unstimulated whole saliva samples will be collected using the passive drool technique at the following time points: 1) immediately following completion of baseline surveys, 2) immediately following the experimental writing task, 3) 1-minute post-cold pressor test, and 4) 10-minutes post-cold pressor test.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Deichert, PhD, Principal Investigator — Black Hills State University
Locations (1):
- Black Hills State University, Spearfish, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
All IPD that underlie results will be in a publication.